CLINICAL TRIAL: NCT05939466
Title: Is Low Dosage of Medical Cannabis Effective for Treating Pain Related to Fibromyalgia?
Brief Title: Medical Cannabis for Treating Pain Related to Fibromyalgia
Acronym: Bedrocan®-LD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universita degli Studi della Basilicata (Other)
Collaborators: San Carlo Public Hospital, Potenza, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PzAOR San Carlo - Bedrocan®
Record Dates: First submitted 2023-06-22; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Medical cannabis; Bedrocan®; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Dronabinol; Medical Marijuana

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FM patients treated with Bedrocan® (Experimental): Medical cannabis was administered by herbal tea or decoction as described by the Ministry of Health through the Ministerial Decree of 9 November 2015.
  Interventions: Drug: Bedrocan®-type cannabis (22% THC, <1% CBD)

INTERVENTIONS:
Drug: Bedrocan®-type cannabis (22% THC, <1% CBD) — Decoction with 100 mg of Bedrocan®-type cannabis (22% THC, <1% CBD)
  Other Names: Medical Cannabis

SUMMARY:
The goal of this interventional study is to learn about the effect of Medicinal Cannabis (Bedrocan®) on Fibromyalgia patients with pain resistant to conventional therapy. The main question the trial aims to answer are:

* Is Bedrocan® effective for treating fibromyalgia-related pain in patients resistant to conventional therapy?
* Can a low dosage of medical cannabis taken as a decoction reduce fibromyalgic pain?

All patients were trained on how to make the decoction: therapy was started with 100 mg/day (1 folder) and increased to 200 mg/day (2 folders) in non-responders.

DETAILED DESCRIPTION:
The study took place in the pain therapy unit of San Carlo Hospital (Potenza, Italy) between March 2021 and September 2021. Over this period, 44 subjects visited the pain unit and underwent specialist evaluation. Fibromyalgia syndrome was confirmed using the Widespread Pain Index (WPI) and Symptom Severity (SS) scale criteria, resulting in the recruitment of 34 subjects. Two participants discontinued therapy due to side effects, while 2 other patients were excluded for not initiating treatment within the required timeframe. Therefore, the final number of recruited fibromyalgic subjects for the study was 30. Among these subjects, those who provided informed written consent for starting the trial with medical cannabis were prescribed Bedrocan® once a month, with a total of 30 prescriptions per month for a duration of 6 months.

All patients were instructed on how to prepare the decoction; the therapy was started with 100 mg/day (1 chart) and increased to 200 mg/day (2 charts) in non-responsive subjects.

The Numerical Rating Scale (NRS) and SF-12 Short Form health questionnaire were used to evaluate pain intensity and the quality of life at the beginning of the study and 6th-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent;
* Age >18 years old;
* Diagnosis of FM confirmed by a rheumatologist;
* Persistent pain symptoms for at least three months without complaints that may otherwise explain the pain condition;
* Persistent pain syndrome on conventional therapy with opioids or non-steroidal anti- inflammatory drugs
* Not having taken medical cannabis in the previous year since the start of the study
* Stopping drug therapy during the trial with cannabis (Bedrocan®).

Exclusion Criteria:

* Specific contraindications to cannabinoid use;
* Pain syndrome not associated with FM
* Major comorbidities like renal impairment, severe liver disease, chronic hepatitis C, history of alcohol or drug addiction
* The presence of cognitive deficits that could impair understanding of the study, completion of questionnaires, or adherence to therapy.
* Pregnant or planning pregnancy women and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 6 months
  Pain intensity evaluated with the Numerical Rating Scale (NRS). NRS involves asking individuals to rate their pain on a numerical scale typically ranging from 0 to 10, where 0 represents no pain and 10 represents the worst possible pain.
Physical state | 6 months
  Physical state was evaluated with the Physical Component Summary of the Short-form health survey SF-12 questionnaire (PCS-12). The PCS-12 provides a summary score that reflects the individual's overall physical health status; it can range from 10.5 to 69.7, with higher scores indicating better physical functioning and well-being.
Mental state | 6 months
  Mental state was evaluated with the Mental Component Summary of the SF-12 questionnaire (MCS-12). MCS-12 provides a summary score, ranging between 7.4 to 72.1, that reflects the individual's overall mental health status. Higher scores on the MCS-12 indicate better mental well-being, while lower scores may indicate higher levels of psychological distress or impairment in social and emotional functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Giardina, Study Director — San Carlo Hospital, Potenza, Italy; Rocco Palmieri, Principal Investigator — San Carlo Hospital, Potenza, Italy
Locations (1):
- Pain Therapy Unit, San Carlo Hospital, Potenza, Italy

IPD SHARING:
Plan to Share IPD: No